CLINICAL TRIAL: NCT00134199
Title: A 6-Month, Randomized, Double-Blind, Placebo And Positive-Controlled Phase 2b Study To Evaluate The Effect Of Various Doses Of CP-945,598 On Weight Loss In Obese Subjects
Brief Title: A Study Of 6-Month Duration To Evaluate The Weight Loss Effect Of Various Doses Of CP-945,598 In Obese Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5351013
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2006-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine

INTERVENTIONS:
Drug: CP-945,598
Drug: sibutramine

SUMMARY:
To evaluate the effect of 6-month administration of CP-945,598 on:

* weight loss and waist circumference,
* blood pressure, cholesterol, glucose
* other biochemical variables like insulin, leptin, ghrelin, adiponectin, PAI 1, TNF-Î± and hsCRP
* the relationship between the concentration of the drug on the blood and the above parameters
* physical and psychosocial functioning, weight related symptoms, treatment satisfaction, appetite/hunger/satiety/craving and mood, anxiety, anhedonia and depression

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects without clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12 lead ECG and clinical laboratory tests
* Body Mass Index (BMI) Â³30 and <40 kg/m2, for subjects with no additional
* co morbidities; BMI Â³27 kg/m2 and <40 kg/m2, for subjects with co morbidities [history of essential hypertension and/or dyslipidemia defined as high LDL (Â³160 mg/dL) or high total cholesterol (Â³240 mg/dL)];

Exclusion Criteria:

* Subjects with resting sitting systolic blood pressure of 140 mmHg or greater or diastolic blood pressure of 90 mmHg or greater.
* Subjects with type 2 diabetes or fasting blood glucose concentration Â³126 mg/dL;
* Subjects with a history of eating disorders like anorexia nervosa or bulimia nervosa
* Subjects on prescription and non-prescription appetite or weight modifying drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2005-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Determine the effect of various doses of CP 945,598 on body weight in obese subjects after 24 weeks of dosing

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of CP 945,598 in a 26 week outpatient setting;; -Explore the effect of CP 945,598 on: waist circumference, PD measurements of selected biochemical variables related to energy deficit and weight loss includ

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Tacoma, Washington